CLINICAL TRIAL: NCT02028507
Title: Phase III Study of Palbociclib in Combination With Exemestane or Fulvestrant vs. Chemotherapy (Capecitabine) in Hormonal Receptor Positive/HER2 Negative Metastatic Breast Cancer Patients With Resistance to Aromatase Inhibitors
Brief Title: Phase III Palbociclib With Endocrine Therapy vs. Capecitabine in HR+/HER2- MBC With Resistance to Aromatase Inhibitors
Acronym: PEARL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Pfizer (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM/2013-02; 2013-003170-27 (EudraCT Number)
Record Dates: First submitted 2014-01-02; First posted 2014-01-07 (Estimated); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Breast Cancer
Keywords: Palbociclib; Capecitabine; Hormonal Receptor positive; HER2 negative; Metastatic Breast Cancer; Resistance to non-steroidal Aromatase inhibitors; Fulvestrant; Exemestane; Aromatase inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Capecitabine; exemestane; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1: Palbociclib plus Exemestane (Experimental): - Cohort 1:Palbociclib 125 mg orally once daily on Day 1 to Day 21 followed by 7 days off treatment on every 28 days cycles in combination with Exemestane 25 mg orally once daily.
  Interventions: Drug: Palbociclib; Drug: Exemestane
- Cohort 1:Capecitabine (Active Comparator): Cohort 1: Capecitabine, 1,250 mg/m2 twice daily for 2 weeks followed by a 1 week rest period, given as 3 weeks cycles. Capecitabine must be administered at a dose of 1,000 mg/m2 twice daily for 2 weeks followed by a 1 week of rest period, given as 3 weeks cycles, in patients over 70 years of age.
  Interventions: Drug: Capecitabine
- Cohort 2: Palbociclib plus Fulvestrant (Experimental): - Cohort 2: Palbociclib 125 mg orally once daily on Day 1 to Day 21 followed by 7 days off treatment on every 28 days cycles in combination with Fulvestrant 500 mg on Days 1 and 15 of Cycle 1, and Day 1 of each subsequent 28 days Cycle.
  Interventions: Drug: Palbociclib; Drug: Fulvestrant
- Cohort 2:Capecitabine (Active Comparator): Cohort 2:Capecitabine, 1,250 mg/m2 twice daily for 2 weeks followed by a 1 week rest period, given as 3 weeks cycles. Capecitabine must be administered at a dose of 1,000 mg/m2 twice daily for 2 weeks followed by a 1 week of rest period, given as 3 weeks cycles, in patients over 70 years of age.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Palbociclib
  Other Names: Ibrance
  Arms: Cohort 1: Palbociclib plus Exemestane; Cohort 2: Palbociclib plus Fulvestrant
Drug: Capecitabine
  Other Names: Xeloda
  Arms: Cohort 1:Capecitabine; Cohort 2:Capecitabine
Drug: Exemestane
  Other Names: aromasil
  Arms: Cohort 1: Palbociclib plus Exemestane
Drug: Fulvestrant
  Other Names: faslodex
  Arms: Cohort 2: Palbociclib plus Fulvestrant

SUMMARY:
This is an international (4 countries) randomized phase III study with 2 cohorts, patients will be randomized 1:1 to endocrine therapy (cohort 1: exemestane 25 mg daily, cohort 2: fulvestrant 500mg days 1 and 15 cycle 1 and then day 1 every 4 weeks) plus palbociclib (125 mg daily x3 weeks every 4 weeks) vs. capecitabine (1,250 mg/m2 twice daily x2 weeks every 3 weeks). Postmenopausal patients with HR+/HER2 MBC are eligible if resistant to previous nonsteroidal aromatase inhibitors (NSAI) (letrozole or anastrozole) in cohort 1 or previous aromatase inhibitors (AI) (letrozole, anastrozole or exemestane) in cohort 2 defined as: recurrence while on or within 12 months after the end of adjuvant treatment with NSAI/AI or progression while on or within 1 month after the end of treatment with NSAI/AI for MBC. Previous chemotherapy is permitted either in the (neo)adjuvant setting and/or as first line for MBC. Patients must have measurable disease according to RECIST 1.1 or bone lesions, lytic or mixed, in the absence of measurable disease.

DETAILED DESCRIPTION:
296 patients have been randomized 1:1 between the experimental arm (Arm A: approximately 125 patients treated with palbociclib plus exemestane) and the control arm (Arm B: approximately 125 patients treated with capecitabine) before the approval of this protocol version (Cohort 1).

Approximately 300 patients will be randomized 1:1 between the experimental arm (Arm A: approximately 150 patients treated with palbociclib plus fulvestrant) and the control arm (Arm B: approximately 150 patients treated with capecitabine) from the approval of this protocol version (Cohort 2).

ELIGIBILITY:
Inclusion Criteria:

1. The patient has signed the informed consent document.
2. a) Patients in cohort 1: Females with histologically confirmed MBC whose disease is resistant to previous non-steroidal aromatase inhibitors (letrozole or anastrozole) b) Patients in cohort 2: Females with histologically confirmed MBC whose disease was resistant to previous aromatase inhibitors (exemestane, letrozole or anastrozole).

   Resistance is defined as: Recurrence while on or within 12 months after the end of adjuvant treatment with NSAI/AI or Progression while on or within 1 month after the end of treatment with NSAI/AI for advanced disease.
3. Previous chemotherapy is permitted either in the (neo) adjuvant setting and/or first line therapy for MBC (chemotherapy administered as "second adjuvant therapy" for locoregional recurrence should be considered as first line chemotherapy for MBC).
4. It is not mandatory to have exemestane, letrozole or anastrozole as the most recent treatment before randomization but recurrence or progression of breast cancer while receiving (or immediately after the enf of) the most recent systemic therapy has to be documented before randomization.
5. Hormonal receptor positive (HR+) breast cancer based on local laboratory determination. HR+ defined as major or equal to 1 percent positive cells by Immunohistochemistry (IHC) for ER and/or Progesterone Receptor (PgR).
6. Documented HER2 negative breast cancer based on local laboratory determination on most recent tumor biopsy. HER2 negative tumor is determined as IHC score 0 or 1+ or negative by ISH (FISH/Chromogenic In Situ Hybridization (CISH)/SISH) defined as a HER2/CEP17 ratio minor to 2 or for single probe assessment a HER2 copy number minor to 4.
7. Measurable disease or at least one bone lesion, lytic or mixed (lytic+blastic), which has not been previously irradiated and is assessable by CT/MRI in the absence of measurable disease according to RECIST 1.1 criteria.
8. Patient is at least 18 years of age.
9. Eastern Cooperative Oncology Group (ECOG) Performance Status minor or equal to 1.
10. Life expectancy major or equal to 12 weeks.
11. Adequate organ and bone marrow function.
12. Postmenopausal women defined as women with:

    Prior bilateral surgical oophorectomy, or Age > 60 years, or Age < 60 years and medically confirmed post-menopausal status defined as spontaneous cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause or follicle-stimulating hormone (FSH) and estradiol blood levels in their respective postmenopausal ranges
13. Resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures to NCI CTCAE version 4.0 Grade minor or equal to 1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator´s discretion).
14. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Have received more than 1 prior chemotherapy regimen for MBC. (NOTE: Chemotherapy administered as "second adjuvant therapy" for locoregional recurrence should be considered one prior chemotherapy for MBC).Other previous anticancer endocrine treatments for advanced disease are allowed.
2. Patients with advanced, symptomatic, visceral spread that are at risk of life-threatening complications in the short term (including patients with massive uncontrolled effusions (pleural, pericardial, peritoneal), pulmonary lymphangitis and over 50% liver involvement).
3. Known active uncontrolled or symptomatic central nervous system (CNS) metastases, carcinomatous meningitis or leptomeningeal disease as indicated by clinical symptoms, cerebral edema, and/or progressive growth. Patients with a history of CNS metastases or cord compression are eligible if they have been definitively treated with local therapy (eg, radiotherapy,) and are clinically stable off anticonvulsants and steroids for at least 4 weeks before randomization.
4. Prior treatment with any CDK4/6, mTOR or PI3K inhibitor (any agent whose mechanism of action is to inhibit the PI3 kinase-mTOR pathway) or capecitabine.
5. a) Patients included in cohort 1: Prior treatment with exemestane in the metastatic setting. If the patient has received exemestane in the adjuvant setting and developed MBC, she will be eligible for the study provided:

   * She has received letrozole/anastrozole as first-line MBC and progressed.
   * At least 1 year has elapsed since the end of adjuvant exemestane treatment. b) Patients included in Cohort 2: Prior treatment with fulvestrant in the metastatic setting. If the patient has received fulvestrant in the adjuvant setting and developed MBC, she will be eligible for the study provided:
   * She has received letrozole/anastrozole as first-line MBC and progressed.
   * At least 1 year has elapsed since the end of adjuvant fulvestrant treatment.
6. Patients treated within the last 7 days prior to randomization with:

   * Food or drugs that are known to be CYP3A4 inhibitors
   * Drugs that are known to be CYP3A4 inducers
   * Drugs that are known to prolong the QT interval
7. Patients who received before randomization:

   * Any investigational agent within 4 weeks
   * Chemotherapy within a period of time that is minor than the cycle length used for that treatment (e.g. less 3 weeks for fluorouracil, doxorubicine, epirubicin or less than 1 week for weekly chemotherapy)
   * Previous endocrine therapy is permitted without any window
   * Radiotherapy within 2 weeks (all acute toxic effects must be resolved to NCI CTCAE version 4.0 grade minor 1, except toxicities not considered a safety risk for the patient at investigator´s discretion) but patients who received prior radiotherapy to less than 25 per cent of bone marrow are not eligible independent of when it was received
   * Major surgery or other anti-cancer therapy not previously specified within 4 weeks, (all acute toxic effects must be resolved to NCI CTCAE version 4.0 grade minor 1, except toxicities not considered a safety risk for the patient at investigator´s discretion)
8. Diagnosis of any other malignancy within 3 years prior to randomization, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix.
9. QTc major 480msec, family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsade de Pointes (TdP).
10. Uncontrolled electrolyte disorders that can compound the effects of a QTc-prolonging drug (eg, hypocalcemia, hypokalemia, hypomagnesemia).
11. Any of the following within 6 months of randomization: myocardial infarction, severe/unstable angina, ongoing cardiac dysrhythmias of NCI CTCAE version 4.0 Grade major or equal to 2, atrial fibrillation of any grade, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident including transient ischemic attack, or symptomatic pulmonary embolism.
12. Difficulties to swallow tablets, malabsorption syndrome disease significantly affecting gastrointestinal function, resection of the stomach or small bowel, or active inflammatory bowel disease or chronic diarrhea.
13. Known hypersensitivity to exemestane, palbociclib, capecitabine, fulvestrant or any of their excipients.
14. Any of the following contraindications for chemotherapy with capecitabine:

    * Known deficiency or family history of deficiency of dihydropyrimidine dehydrogenase.
    * Requirement for concurrent use of the antiviral agent sorivudine (antiviral) or chemically related analogues, such as brivudine.
15. Only for patients in Cohort 2 any of the following contraindications for treatment with fulvestrant:

    - Bleeding diathesis (i.e., disseminated intravascular coagulation, clotting factor deficiency) or long-term anticoagulant therapy (other than antiplatelet therapy and low dose warfarin) provided that the International Normalised Ratio (INR) is less than 1.6.
16. Known human immunodeficiency virus infection.
17. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
18. Recent or active suicidal ideation or behavior

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 693 (Actual)
Dates: Start 2014-03-13 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2021-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — IiSGM, Universidad Complutense de Madrid, Madrid, Spain.
Locations (37):
- Austria (3):
  - Universitätsklinik für Innere Medizin III, Salzburg
  - Landes-Krankenhaus Steyr, Steyr
  - Universitätsklinik für Innere Medizin I, Vienna
- Hungary (5):
  - Semmelweis Egyetem, Budapest
  - Szent Imre Egyetemi Oktatókórház, Budapest
  - National Institute of Oncology, Budapest
  - Onkotherápiás Klinika, Szeged
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház-Rendelőintézet, Szolnok
- Israel (4):
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Spain (25):
  - ICO de L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Centro Oncológico de Galicia, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario Germans Trias i Pujol, Barcelona
  - Hospital San Pedro De Alcántara, Cáceres
  - Complejo Hospitalario Universitario Reina Sofía, Córdoba
  - Hospital de Donostia, Donostia / San Sebastian
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital de León, León
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Clínico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Virgen de La Salud, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario La Fe, Valencia
  - Hospital Clínico Universitario de Zaragoza "Lozano Blesa", Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Martin M, Zielinski C, Ruiz-Borrego M, Carrasco E, Turner N, Ciruelos EM, Munoz M, Bermejo B, Margeli M, Anton A, Kahan Z, Csoszi T, Casas MI, Murillo L, Morales S, Alba E, Gal-Yam E, Guerrero-Zotano A, Calvo L, de la Haba-Rodriguez J, Ramos M, Alvarez I, Garcia-Palomo A, Huang Bartlett C, Koehler M, Caballero R, Corsaro M, Huang X, Garcia-Saenz JA, Chacon JI, Swift C, Thallinger C, Gil-Gil M. Palbociclib in combination with endocrine therapy versus capecitabine in hormonal receptor-positive, human epidermal growth factor 2-negative, aromatase inhibitor-resistant metastatic breast cancer: a phase III randomised controlled trial-PEARL. Ann Oncol. 2021 Apr;32(4):488-499. doi: 10.1016/j.annonc.2020.12.013. Epub 2020 Dec 29. PMID 33385521
- [Result] Martin M, Zielinski C, Ruiz-Borrego M, Carrasco E, Ciruelos EM, Munoz M, Bermejo B, Margeli M, Csoszi T, Anton A, Turner N, Casas MI, Morales S, Alba E, Calvo L, de la Haba-Rodriguez J, Ramos M, Murillo L, Santaballa A, Alonso-Romero JL, Sanchez-Rovira P, Corsaro M, Huang X, Thallinger C, Kahan Z, Gil-Gil M. Overall survival with palbociclib plus endocrine therapy versus capecitabine in postmenopausal patients with hormone receptor-positive, HER2-negative metastatic breast cancer in the PEARL study. Eur J Cancer. 2022 Jun;168:12-24. doi: 10.1016/j.ejca.2022.03.006. Epub 2022 Apr 13. PMID 35429901
- [Result] Kahan Z, Gil-Gil M, Ruiz-Borrego M, Carrasco E, Ciruelos E, Munoz M, Bermejo B, Margeli M, Anton A, Casas M, Csoszi T, Murillo L, Morales S, Calvo L, Lang I, Alba E, de la Haba-Rodriguez J, Ramos M, Lopez IA, Gal-Yam E, Garcia-Palomo A, Alvarez E, Gonzalez-Santiago S, Rodriguez CA, Servitja S, Corsaro M, Rodrigalvarez G, Zielinski C, Martin M. Health-related quality of life with palbociclib plus endocrine therapy versus capecitabine in postmenopausal patients with hormone receptor-positive metastatic breast cancer: Patient-reported outcomes in the PEARL study. Eur J Cancer. 2021 Oct;156:70-82. doi: 10.1016/j.ejca.2021.07.004. Epub 2021 Aug 20. PMID 34425406
- [Result] Guerrero-Zotano A, Belli S, Zielinski C, Gil-Gil M, Fernandez-Serra A, Ruiz-Borrego M, Ciruelos Gil EM, Pascual J, Munoz-Mateu M, Bermejo B, Margeli Vila M, Anton A, Murillo L, Nissenbaum B, Liu Y, Herranz J, Fernandez-Garcia D, Caballero R, Lopez-Guerrero JA, Bianco R, Formisano L, Turner N, Martin M. CCNE1 and PLK1 Mediate Resistance to Palbociclib in HR+/HER2- Metastatic Breast Cancer. Clin Cancer Res. 2023 Apr 14;29(8):1557-1568. doi: 10.1158/1078-0432.CCR-22-2206. PMID 36749874
- See also: GEICAM is a Spanish Breast Cancer Research Group — http://www.geicam.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 92 patients were screening failure. A total of 601 patients were included in this study from March 2014 to July 2018. Cohort 1 included 296 patients (153 on palbociclib plus exemestane and 143 on capecitabine) and cohort 2 included 305 patients (149 on palbociclib plus fulvestrant and 156 on capecitabine).
Groups:
- Cohort 1: Palbociclib Plus Exemestane: Cohort 1: Palbociclib 125 mg orally once daily on Day 1 to Day 21 followed by 7 days off treatment on every 28 days cycles in combination with Exemestane 25 mg orally once daily.
  Palbociclib
  Exemestane
- Cohort 1: Capecitabine: Cohort 1: Capecitabine, 1,250 mg/m2 twice daily for 2 weeks followed by a 1 week rest period, given as 3 weeks cycles. Capecitabine must be administered at a dose of 1,000 mg/m2 twice daily for 2 weeks followed by a 1 week of rest period, given as 3 weeks cycles, in patients over 70 years of age.
  Capecitabine
- Cohort 2: Palbociclib Plus Fulvestrant: Cohort 2: Palbociclib 125 mg orally once daily on Day 1 to Day 21 followed by 7 days off treatment on every 28 days cycles in combination with Fulvestrant 500 mg on Days 1 and 15 of Cycle 1, and Day 1 of each subsequent 28 days Cycle.
  Palbociclib
  Fulvestrant
- Cohort 2: Capecitabine: Cohort 2: Capecitabine, 1,250 mg/m2 twice daily for 2 weeks followed by a 1 week rest period, given as 3 weeks cycles. Capecitabine must be administered at a dose of 1,000 mg/m2 twice daily for 2 weeks followed by a 1 week of rest period, given as 3 weeks cycles, in patients over 70 years of age.
  Capecitabine
Period: Overall Study
Arm/Group | Cohort 1: Palbociclib Plus Exemestane | Cohort 1: Capecitabine | Cohort 2: Palbociclib Plus Fulvestrant | Cohort 2: Capecitabine
Started | 153 | 143 | 149 | 156
Completed | 0 | 0 | 0 | 0
Not Completed | 153 | 143 | 149 | 156
Not completed — Progressive Disease | 122 | 90 | 102 | 89
Not completed — Adverse Event | 8 | 25 | 3 | 16
Not completed — Withdrawal by Subject | 6 | 8 | 5 | 9
Not completed — Protocol Violation | 2 | 4 | 1 | 3
Not completed — Physician Decision | 0 | 4 | 0 | 0
Not completed — Death | 1 | 0 | 1 | 3
Not completed — Patient Required Therapy/Procedure Not Permitted | 0 | 1 | 0 | 1
Not completed — Second Invasive Primary Malignancy | 1 | 0 | 0 | 1
Not completed — Randomized But Not Treated | 3 | 6 | 0 | 4
Not completed — Enzyme defect | 0 | 0 | 0 | 1
Not completed — Patient was not able to take whole dose of capecitabine | 0 | 0 | 0 | 1
Not completed — Ongoing at date of cut-off 30-May-2019 | 10 | 5 | 37 | 28

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Palbociclib Plus Exemestane: - Cohort 1:Palbociclib 125 mg orally once daily on Day 1 to Day 21 followed by 7 days off treatment on every 28 days cycles in combination with Exemestane 25 mg orally once daily.
  Palbociclib
  Exemestane
- Cohort 1:Capecitabine: Cohort 1: Capecitabine, 1,250 mg/m2 twice daily for 2 weeks followed by a 1 week rest period, given as 3 weeks cycles. Capecitabine must be administered at a dose of 1,000 mg/m2 twice daily for 2 weeks followed by a 1 week of rest period, given as 3 weeks cycles, in patients over 70 years of age.
  Capecitabine
- Cohort 2: Palbociclib Plus Fulvestrant: - Cohort 2: Palbociclib 125 mg orally once daily on Day 1 to Day 21 followed by 7 days off treatment on every 28 days cycles in combination with Fulvestrant 500 mg on Days 1 and 15 of Cycle 1, and Day 1 of each subsequent 28 days Cycle.
  Palbociclib
  Fulvestrant
- Cohort 2:Capecitabine: Cohort 2:Capecitabine, 1,250 mg/m2 twice daily for 2 weeks followed by a 1 week rest period, given as 3 weeks cycles. Capecitabine must be administered at a dose of 1,000 mg/m2 twice daily for 2 weeks followed by a 1 week of rest period, given as 3 weeks cycles, in patients over 70 years of age.
  Capecitabine
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Palbociclib Plus Exemestane | Cohort 1:Capecitabine | Cohort 2: Palbociclib Plus Fulvestrant | Cohort 2:Capecitabine | Total
Number analyzed (Participants) | 153 | 143 | 149 | 156 | 601
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 97 | 98 | 93 | 103 | 391
  >=65 years | 56 | 45 | 56 | 53 | 210
Age, Continuous [Median (Full Range); unit: years] | 60 [31 to 89] | 60 [38 to 87] | 62 [38 to 86] | 60 [33 to 85] | 60 [31 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 143 | 149 | 156 | 601
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic Or Latino | 20 | 21 | 16 | 18 | 75
  Not Hispanic Or Latino | 128 | 118 | 129 | 136 | 511
  Unknown | 5 | 4 | 4 | 2 | 15
Region of Enrollment [Number; unit: participants]
  Austria | 5 | 1 | 4 | 5 | 15
  Hungary | 10 | 8 | 22 | 19 | 59
  Israel | 7 | 6 | 12 | 14 | 39
  Spain | 131 | 128 | 111 | 118 | 488
Eastern Cooperative Oncology Group (ECOG) status [Count of Participants; unit: Participants] — ECOG score runs from 0 to 5, with 0 denoting perfect health and 5 death. 0 - Asymptomatic
  1. - Symptomatic but completely ambulatory
  2. - Symptomatic, <50% in bed during the day
  3. - Symptomatic, >50% in bed, but not bedbound
  4. - Bedbound
  5. - Death
  Participants
    ECOG 0 | 85 | 84 | 90 | 93 | 352
    ECOG 1 | 68 | 59 | 59 | 63 | 249
Visceral disease [Count of Participants; unit: Participants]
  Yes | 103 | 94 | 97 | 102 | 396
  No | 50 | 48 | 52 | 54 | 204
  Not available | 0 | 1 | 0 | 0 | 1
Hormone receptor status [Count of Participants; unit: Participants]
  Estrogen-receptor (ER) positive and progesterone-receptor (PR) positive | 114 | 103 | 114 | 118 | 449
  ER positive and PR negative | 36 | 38 | 33 | 33 | 140
  ER negative and PR positive or ER positive and PR not available | 2 | 2 | 2 | 5 | 11
  Triple negative | 1 | 0 | 0 | 0 | 1
ESR1 mutational status [Count of Participants; unit: Participants]
  Wild-type | 104 | 89 | 102 | 98 | 393
  Mutant | 41 | 37 | 38 | 48 | 164
  Not available | 8 | 17 | 9 | 10 | 44
Sensitivity to prior endocrine therapy [Count of Participants; unit: Participants]
  Yes | 107 | 104 | 119 | 122 | 452
  No | 46 | 39 | 30 | 34 | 149
Number of prior lines of endocrine therapy for metastatic breast cancer (MBC) [Count of Participants; unit: Participants]
  No prior endocrine therapy for MBC | 30 | 31 | 38 | 44 | 143
  1 | 82 | 70 | 85 | 90 | 327
  2 | 35 | 34 | 12 | 9 | 90
  3 | 3 | 4 | 1 | 1 | 9
  Maintenance after chemotherapy | 3 | 4 | 12 | 12 | 31
  Combination | 0 | 0 | 1 | 0 | 1
Prior chemotherapy for MBC [Count of Participants; unit: Participants]
  Yes | 48 | 41 | 41 | 41 | 171
  No | 105 | 102 | 108 | 115 | 430
Line at study entry [Count of Participants; unit: Participants]
  1st line | 27 | 31 | 38 | 43 | 139
  2nd line | 63 | 50 | 76 | 79 | 268
  ≥3rd line | 63 | 62 | 35 | 34 | 194
Status at initial diagnosis [Count of Participants; unit: Participants]
  M0: Cancer has not spread to other parts of the body | 127 | 109 | 115 | 120 | 471
  M1: Cancer has spread to other parts of the body | 26 | 34 | 34 | 36 | 130
Histopathology type [Count of Participants; unit: Participants]
  Breast Invasive Ductal Carcinoma | 122 | 117 | 117 | 125 | 481
  Breast Invasive Lobular Carcinoma | 23 | 24 | 24 | 20 | 91
  Other | 3 | 1 | 4 | 8 | 16
  Not Available/Not Done | 5 | 1 | 4 | 3 | 13
Histologic grade [Count of Participants; unit: Participants] — Cancer cells are given a Grade (G) when they are removed from the breast and checked under a microscope. The G is based on how much the cancer cells look like normal cells.
  G1 or well differentiated (score 3, 4, or 5): cells are slower-growing, and look more like normal breast tissue.
  G2 or moderately differentiated (score 6, 7): cells are growing at a speed of and look like cells somewhere between G1 and 3.
  G3 or poorly differentiated (score 8, 9): cells look very different from normal and will probably grow and spread faster.
  Participants
    G1, Well Differentiated | 17 | 15 | 13 | 14 | 59
    G2, Moderately Differentiated | 68 | 57 | 70 | 72 | 267
    G3, Poorly Differentiated | 36 | 37 | 38 | 40 | 151
    GX, Unknown | 23 | 23 | 19 | 19 | 84
    Not Available/Not Done | 9 | 11 | 9 | 11 | 40

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: The primary efficacy variable is PFS based on the investigator's assessment. PFS is defined as the time from randomization to the first documented progressive disease based on the investigator's assessment, using RECIST version 1.1, or death from any cause, whichever occurs first.
  Estrogen Receptor 1 (ESR1) mutational status will be determined in circulating free DNA (cDNA) obtained from.
  Disease assessments will be performed at baseline and every 8 weeks (± 7 days) from the start of treatment and every 12 weeks (±7 days) after 120 weeks of treatment baseline plasma samples and will be prospectively determined before the interims or final analyses. ESR1 mutational status will be blinded to the patients, investigators and study team.
Time Frame: Through study treatment, and average of 8 months
Population: The Intent to treat population (ITT) include all patients who were randomized, with study drug/medication assignment designated according to initial randomization.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Cohort 1: Palbociclib Plus Exemestane | Cohort 1: Capecitabine | Cohort 2: Palbociclib Plus Fulvestrant | Cohort 2: Capecitabine
Number analyzed (Participants) | 153 | 143 | 149 | 156
month | 7.3 [5.6 to 9.7] | 9.4 [7.4 to 11.8] | 7.5 [5.7 to 10.9] | 10 [6.3 to 12.9]

2. Secondary Outcome: PFS Estrogen Receptor 1 (ESR1) Wild Type
Description: PFS is defined as the time from randomization to the first documented progressive disease based on the investigator's assessment, using RECIST version 1.1, or death from any cause, whichever occurs first. PFS data will be censored on the date of the last tumor assessment on study for patients who do not have objective tumor progression and who do not die while on study. Patients lacking an evaluation of tumor response after randomization will have their PFS time censored on the date of randomization with 1 day duration. Additionally, patients who start a new anti-cancer therapy prior to documented PD will be censored at the date of the last tumor assessment prior to the start of the new therapy.
Time Frame: From randomization date to date of first documentation of progression or death (an average of 8 months)
Population: ESR1 wild type population include patients with ESR1 mutational status as wild type at study entry.
  * Exemestane or Fulvestrant plus Palbociclib ESR1 wild type population: Cohort 1 (n=153) of which ESR1 wild type (n=104) and cohort 2 (n=149) of which ESR1 wild type (n=102). Total ESR1 wild type 206
  * Capecitabine ESR1 wild type population: Cohort 1 (n=143) of which ESR1 wild type (n=89) and cohort 2 (n=156) of which ESR1 wild type (n=98). Total ESR1 wild type 187
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Exemestane or Fulvestrant Plus Palbociclib ESR1 Wild Type Population; Capecitabine ESR1 Wild Type Population: The ESR1 wild type population will include all patients who are randomized, with study drug/medication assignment designated according to initial randomization and whose tumor had estrogen receptor (ESR1) mutational status as wild type at study entry.
Arm/Group | Exemestane or Fulvestrant Plus Palbociclib ESR1 Wild Type Population | Capecitabine ESR1 Wild Type Population
Number analyzed (Participants) | 206 | 187
months | 8.0 [6.5 to 10.9] | 10.6 [7.4 to 13.0]

3. Secondary Outcome: Overall Survival (OS) ESR1 Wild Type
Description: OS is defined as the time from the date of randomization to the date of death from any cause.
Time Frame: From randomization until death (up to approximately 34 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Exemestane or Fulvestrant Plus Palbociclib ESR1 Wild Type Population | Capecitabine ESR1 Wild Type Population
Number analyzed (Participants) | 206 | 187
months | 33.7 [27.6 to 45.1] | 32 [28 to 46.9]

4. Secondary Outcome: Objective Response Rate (ORR) ESR1 Wild Type
Description: Complete Response (CR) plus Partial Response (PR) based on the investigator's assessment according to the RECIST version 1.1 in patients randomized with measurable disease.
  Tumor assessment will be performed at baseline, the same method of measurement used at baseline will be used for further evaluations, that will be conducted every 8 weeks (±7days). The best response across treatment will be recorded. OR is defined as the complete plus partial responses out of the patients who had measurable disease at baseline.
Time Frame: Through study treatment, and average of 8 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Exemestane or Fulvestrant Plus Palbociclib ESR1 Wild Type Population | Capecitabine ESR1 Wild Type Population
Number analyzed (Participants) | 206 | 187
Participants | 47 | 55

5. Secondary Outcome: Clinical Benefit Rate (CBR) ESR1 Wild Type
Description: CB is defined as complete response (CR), partial response (PR), or stable disease (SD) based on the investigator´s assessment lasting more than 24 weeks according to the RECIST version 1.1 in all randomized patients (ITT population). Per RECIST, CR is defined as the disappearance of all target lesions; PR is defined as an >=30% decrease in the sum of the longest diameter of target lesions; SD is defined as a failure to meet criteria for CR or PR in the absence of progressive disease. Overall Response (OR) = CR + PR.
Time Frame: Through study treatment, and average of 8 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Exemestane or Fulvestrant Plus Palbociclib ESR1 Wild Type Population; Capecitabine ESR1 Wild Type Population: The ESR1 wild type population include all patients who are randomized, with study drug/medication assignment designated according to initial randomization and whose tumor had estrogen receptor (ESR1) mutational status as wild type at study entry.
Arm/Group | Exemestane or Fulvestrant Plus Palbociclib ESR1 Wild Type Population | Capecitabine ESR1 Wild Type Population
Number analyzed (Participants) | 206 | 187
Participants | 157 | 154

6. Secondary Outcome: Response Duration (RD) ESR1 Wild Type
Description: Tumor response was assessed using Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) criteria. RD was defined as the time from the first documentation of objective tumor response (complete response (CR) or partial response (PR)) to the first documented progressive disease (PD), or to death due to any cause, whichever occurs first. Per RECIST, CR is defined as the disappearance of all target lesions; PR is defined as an >=30% decrease in the sum of the longest diameter of target lesions; PD is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Through study treatment, and average of 8 months
Population: Safety population includes all patients randomized in the study who received at least one dose of treatment, according to the actual treatment received.
  Patients from Safety Population with Measurable Disease and Best Response Complete or Partial.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Exemestane or Fulvestrant Plus Palbociclib ESR1 Wild Type Population | Capecitabine ESR1 Wild Type Population
Number analyzed (Participants) | 47 | 55
months | 9.7 [8.7 to 21.7] | 11.2 [7.2 to 17.3]

7. Secondary Outcome: The Number of Participants Who Experienced Adverse Events (AE)
Description: Safety will be assessed by standard clinical and laboratory tests (hematology, serum chemistry). Adverse events grade will be defined by the NCI CTCAE v4.0.
  Safety assessments were performed at baseline and during the study: Vital signs (blood pressure, pulse, temperature), Laboratory (hemoglobin, White Blood Cell, Absolute Neutrophils, platelet count, fasting glucose, alkaline phosphatase, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, serum creatinine, sodium, potassium, magnesium, total calcium.
  AEs were graded according to NCI-CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) version 4.03.
Time Frame: Through study treatment, and average of 8 months
Population: Safety population include patients randomized in the study who received at least one dose of treatment, according to the actual treatment received.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 + 2: Capecitabine: Cohort 1 and 2: Capecitabine, 1,250 mg/m2 twice daily for 2 weeks followed by a 1 week rest period, given as 3 weeks cycles. Capecitabine must be administered at a dose of 1,000 mg/m2 twice daily for 2 weeks followed by a 1 week of rest period, given as 3 weeks cycles, in patients over 70 years of age.
  Capecitabine
Arm/Group | Cohort 1: Palbociclib Plus Exemestane | Cohort 2: Palbociclib Plus Fulvestrant | Cohort 1 + 2: Capecitabine
Number analyzed (Participants) | 150 | 149 | 289
Participants | 147 | 148 | 286

8. Secondary Outcome: Overall Change From Baseline Between Treatment Comparison in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Functional Scale Scores
Description: The EORTC QLQ C30 is a 30 item questionnaire composed of functional scales, a global health/quality of life and cancer related symptoms.
  All of the scales and single-item measures range are scored from 0 to 100. A high scale score represents a high / healthy level of functioning.
  Change from baseline has been calculated as each visit score minus baseline score.
  The change from baseline of EORTC QLQ-C30 subscales have been analyzed using linear mixed models, including treatment group, visit, the interaction between treatment group and visit, baseline score and stratification factors as covariates. Overall mean of change and CI 95% has been retrieved from this analysis.
Time Frame: Assessed at Baseline, cycles 3, 5, 7, and then at every 3 cycles until the end of treatment, and at the visit after treatment, an average of 8 months.
Population: QoL population: a subset of enrolled patients with available QoL questionnaires (the baseline and at least one more).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib: * Cohort 1: Palbociclib 125 mg orally once daily on Day 1 to Day 21 followed by 7 days off treatment on every 28 days cycles in combination with Exemestane 25 mg orally once daily.
  * Cohort 2: Palbociclib 125 mg orally once daily on Day 1 to Day 21 followed by 7 days off treatment on every 28 days cycles in combination with Fulvestrant 500 mg on Days 1 and 15 of Cycle 1, and Day 1 of each subsequent 28 days Cycle.
- Cohort 1 and 2: Capecitabine: Capecitabine, 1,250 mg/m2 twice daily for 2 weeks followed by a 1 week rest period, given as 3 weeks cycles. Capecitabine must be administered at a dose of 1,000 mg/m2 twice daily for 2 weeks followed by a 1 week of rest period, given as 3 weeks cycles, in patients over 70 years of age.
  Capecitabine
Arm/Group | Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib | Cohort 1 and 2: Capecitabine
Number analyzed (Participants) | 268 | 269
units on a scale
  Global health status / QoL | 3.28 [1.06 to 5.49] | 1.97 [-0.33 to 4.29]
  Physical functioning | -1.73 [-3.94 to 0.48] | -2.94 [-5.07 to -0.81]
  Role functioning | -1.09 [-4.45 to 2.27] | -4.97 [-7.82 to -2.12]
  Emotional functioning | 6.78 [3.67 to 9.88] | 8.67 [6.04 to 11.29]
  Cognitive functioning | -2.18 [-4.91 to 0.54] | -2.42 [-4.66 to -0.18]
  Social functioning | -0.67 [-3.43 to 2.07] | -3.01 [-5.45 to -0.56]

9. Secondary Outcome: Overall Change From Baseline Between Treatment Comparison in EORTC QLQ-C30 Symptom Scale Scores
Description: The EORTC QLQ C30 is a 30 item questionnaire composed of functional scales, a global health/quality of life and cancer related symptoms.
  All of the scales and single-item measures range are scored from 0 to 100. A high scale score represents a high level of symptomatology / problems.
  Change from baseline has been calculated as each visit score minus baseline score.
  The change from baseline of EORTC QLQ-C30 subscales have been analyzed using linear mixed models, including treatment group, visit, the interaction between treatment group and visit, baseline score and stratification factors as covariates. Overall mean of change and CI 95% has been retrieved from this analysis.
Time Frame: as for outcome 8
Population: QoL population: a subset of enrolled patients with available QoL questionnaires (the baseline and at least one more).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib | Cohort 1 and 2: Capecitabine
Number analyzed (Participants) | 268 | 269
units on a scale
  Fatigue | 3.85 [0.82 to 6.88] | 5.79 [3.14 to 8.43]
  Nausea and vomiting | 1.65 [-0.02 to 3.33] | 1.45 [-0.07 to 2.98]
  Pain | -1.79 [-4.86 to 1.27] | -1.90 [-4.7 to 0.91]
  Dyspnoea | 2.73 [-0.64 to 6.11] | -0.05 [-2.44 to 2.34]
  Insomnia | -3.04 [-6.63 to 0.54] | -5.94 [-8.92 to -2.97]
  Appetite loss | 2.99 [-0.30 to 6.30] | 1.04 [-1.57 to 3.65]
  Constipation | 3.91 [0.56 to 7.27] | -1.45 [-4.10 to 1.19]
  Diarrhoea | 3.67 [1.06 to 6.29] | 6.73 [4.61 to 8.85]
  Financial difficulties | -1.31 [-4.74 to 2.10] | 1.73 [-1.11 to 4.59]

10. Secondary Outcome: Overall Change From Baseline Between Treatment Comparison in European Organization for Research and Treatment of Cancer Breast Cancer Module (EORTC QLQ BR23) Functional Scale Scores
Description: The EORTC QLQ BR23 is a 23 item breast cancer specific companion module to the EORTC QLQ C30 and consists of functional scales and symptom subscales.
  All of the scales and single-item measures range are scored from 0 to 100. A high score for the functional scales represents a high/healthy level of functioning.
  Change from baseline has been calculated as each visit score minus baseline score.
  The change from baseline of EORTC QLQ-BR23 subscales have been analyzed using linear mixed models, including treatment group, visit, the interaction between treatment group and visit, baseline score and stratification factors as covariates. Overall mean of change and CI 95% has been retrieved from this analysis.
Time Frame: as for outcome 8
Population: QoL population: a subset of enrolled patients with available QoL questionnaires (the baseline and at least one more).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib | Cohort 1 and 2: Capecitabine
Number analyzed (Participants) | 268 | 269
units on a scale
  Body image | -1.83 [-4.73 to 1.06] | 0.14 [-2.16 to 2.44]
  Sexual functioning | 2.94 [0.56 to 5.31] | 1.72 [-0.37 to 3.81]
  Sexual enjoyment | -6.32 [-11.86 to -0.78] | -4.32 [-9.25 to 0.60]
  Future perspective | 13.80 [9.61 to 17.99] | 15.22 [11.66 to 18.78]

11. Secondary Outcome: Overall Change From Baseline Between Treatment Comparison in EORTC QLQ BR23 Symptom Scale Scores
Description: The EORTC QLQ BR23 is a 23 item breast cancer specific companion module to the EORTC QLQ C30 and consists of functional scales and symptom subscales.
  All of the scales and single-item measures range are scored from 0 to 100. A high score for the functional scales represents a high level of symptomatology / problems.
  Change from baseline has been calculated as each visit score minus baseline score.
  The change from baseline of EORTC QLQ-BR23 subscales have been analyzed using linear mixed models, including treatment group, visit, the interaction between treatment group and visit, baseline score and stratification factors as covariates. Overall mean of change and CI 95% has been retrieved from this analysis.
Time Frame: as for outcome 8
Population: QoL population: a subset of enrolled patients with available QoL questionnaires (the baseline and at least one more).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib | Cohort 1 and 2: Capecitabine
Number analyzed (Participants) | 268 | 269
units on a scale
  Systemic therapy side effects | 5.61 [3.29 to 7.94] | 4.49 [2.88 to 6.10]
  Breast symptoms | -0.42 [-2.31 to 1.46] | -2.00 [-3.46 to -0.53]
  Arm symptoms | -2.26 [-4.44 to -0.08] | -2.09 [-4.02 to -0.15]
  Upset by hair loss | 8.35 [2.25 to 14.45] | -1.96 [-7.53 to 3.60]

12. Secondary Outcome: Overall Change From Baseline Between Treatment Comparison in EuroQoL 5D (EQ-5D) Health Index Scores
Description: EQ 5D is a 6 item instrument which assess health status in terms of a single index value. Consists of 5 descriptors of current health state (mobility, self-care, usual activities, pain/discomfort, anxiety/depression); patient is asked to rate each state on 3 level scale (1=no problem, 2=some problem, 3=extreme problem). Higher levels indicating greater severity/impairment. It includes a visual analogue scale (EQ VAS) which records patient's self-rated health on a scale from 0 (worst imaginable) to 100 (best imaginable). Published weights allows for the creation of a single summary score. Overall scores range from 0 to 1 (low score=higher level of dysfunction, 1=perfect health).
  The change from baseline of EQ-5D subscales have been analyzed using linear mixed models, including treatment group, visit, the interaction between treatment group and visit, baseline score and stratification factors as covariates. Overall mean of change and CI 95% has been retrieved from this analysis.
Time Frame: Assessed at Baseline, cycles 3, 5, 7, and then at every 3 cycles until the end of treatment, and at the visit after treatment. An average of 8 months, an average of 1 year, and an average of 2 years.
Population: QoL population: a subset of enrolled patients with available QoL questionnaires (the baseline and at least one more).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib | Cohort 1 and 2: Capecitabine
Number analyzed (Participants) | 268 | 269
units on a scale | 0.72 [0.69 to 0.74] | 0.71 [0.69 to 0.73]

13. Secondary Outcome: Overall Change From Baseline Between Treatment Comparison in EQ-5D Visual Analog Scale (VAS) Scores Scale
Description: The EuroQol-5D (version 3L) is a brief self-administered, validated instrument consisting of 2 parts. The second part consists of the EQ-5D general health status as measured by a visual analog scale (EQ-5D VAS). EQ-5D VAS measures the participant's self-rated health status on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state).
  The change from baseline of EQ-5D subscales have been analyzed using linear mixed models, including treatment group, visit, the interaction between treatment group and visit, baseline score and stratification factors as covariates. Overall mean of change and CI 95% has been retrieved from this analysis.
Time Frame: as for outcome 12
Population: QoL population: a subset of enrolled patients with available QoL questionnaires (the baseline and at least one more).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib | Cohort 1 and 2: Capecitabine
Number analyzed (Participants) | 268 | 269
units on a scale | 67.1 [65.3 to 69] | 66.6 [64.9 to 68.2]

14. Secondary Outcome: Time to Deterioration (TTD) in EORTC QLQ-C30 Functional Scale
Description: Time to deterioration is defined as the time from the date of randomization to the date of first detection of deterioration. Deterioration is defined as a change from baseline ≥ minimally important difference (MID) as a change from baseline ≤ -MID for EORTC QLQ-C30 functional scales, global health status/QOL score. Patients without deterioration have been censored at their last quality of life assessment. For patients with no post-baseline assessment time to deterioration have been censored at Day 1.
Time Frame: as for outcome 8
Population: QoL population: a subset of enrolled patients with available QoL questionnaires (the baseline and at least one more).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib | Cohort 1 and 2: Capecitabine
Number analyzed (Participants) | 268 | 269
months
  Global health status/quality of life | 8.3 [6 to 11.1] | 5.3 [4.2 to 8.7]
  Physical functioning | 5.6 [3.7 to 6.9] | 2.8 [1.9 to 3.4]
  Role functioning | 8.3 [5.9 to 11.5] | 4.2 [3 to 5]
  Emotional functioning | 8.5 [5.9 to 12.5] | 11.1 [5.5 to 17.5]
  Cognitive functioning | 11.1 [6.7 to 16.8] | 6.6 [4.9 to 8.8]
  Social functioning | 8.8 [7.1 to 13.1] | 4.4 [3.7 to 6.5]
Statistical Analysis 1: Comparison: Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib vs Cohort 1 and 2: Capecitabine; This statistical Analysis corresponds to Global health status/quality of life scale; Test type: Superiority; p = 0.003, Regression, Cox; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.55 to 0.89]
Statistical Analysis 2: Comparison: Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib vs Cohort 1 and 2: Capecitabine; This statistical Analysis corresponds to Physical functioning scale; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.50 to 0.76]
Statistical Analysis 3: Comparison: Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib vs Cohort 1 and 2: Capecitabine; This statistical Analysis corresponds to Role functioning scale; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.51 to 0.79]
Statistical Analysis 4: Comparison: Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib vs Cohort 1 and 2: Capecitabine; This statistical Analysis corresponds to Emotional functioning scale; Test type: Superiority; p = 0.818, Regression, Cox; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.76 to 1.25]
Statistical Analysis 5: Comparison: Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib vs Cohort 1 and 2: Capecitabine; This statistical Analysis corresponds to Cognitive functioning scale; Test type: Superiority; p = 0.004, Regression, Cox; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.54 to 0.89]
Statistical Analysis 6: Comparison: Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib vs Cohort 1 and 2: Capecitabine; This Statistical Analysis corresponds to Social functioning scale; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.49 to 0.78]

15. Secondary Outcome: Time to Deterioration (TTD) in EORTC QLQ-C30 Symptom Scale
Description: Time to deterioration is defined as the time from the date of randomization to the date of first detection of deterioration. Deterioration is defined as a change from baseline ≥ minimally important difference (MID) for EORTC QLQ-C30 symptom scores. Patients without deterioration have been censored at their last quality of life assessment. For patients with no post-baseline assessment time to deterioration have been censored at Day 1.
  999 means value not estimated.
Time Frame: as for outcome 8
Population: QoL population: a subset of enrolled patients with available QoL questionnaires (the baseline and at least one more). NA (Not Available): the statistical program has not been able to estimate the upper limit of the interval because of the lower number of participants answering the applicable questions.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib | Cohort 1 and 2: Capecitabine
Number analyzed (Participants) | 268 | 269
months
  Fatigue | 3.9 [3.7 to 5.6] | 2.8 [1.9 to 3.1]
  Nausea and vomiting | 17.3 [9.2 to 24.4] | 10 [4.5 to 14.1]
  Pain | 6.2 [5.6 to 11.1] | 6.2 [4.2 to 9.4]
  Dyspnea | 14.8 [11 to 23.2] | 17.8 [12.2 to NA] — NA (Not Available): the statistical program has not been able to estimate the upper limit of the interval because of the lower number of participants answering the applicable questions.
  Insomnia | 14.8 [11.1 to 23.2] | 10.7 [7.5 to 18.2]
  Appetite loss | 17.4 [11.4 to 27.6] | 9.6 [6.5 to 17.7]
  Constipation | 12.4 [8.6 to 18.6] | 16.3 [8.3 to 24.5]
  Diarrhea | 28.1 [13 to NA] — NA (Not Available): the statistical program has not been able to estimate the upper limit of the interval because of the lower number of participants answering the applicable questions. | 4.9 [3.5 to 9.2]
  Financial difficulties | 25.2 [19.4 to NA] — NA (Not Available): the statistical program has not been able to estimate the upper limit of the interval because of the lower number of participants answering the applicable questions. | 19.1 [17.7 to NA] — NA (Not Available): the statistical program has not been able to estimate the upper limit of the interval because of the lower number of participants answering the applicable questions.
Statistical Analysis 1: Comparison: Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib vs Cohort 1 and 2: Capecitabine; This Statistical Analysis corresponds to Fatigue scale; Test type: Superiority; p = 0.001, Regression, Cox; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.57 to 0.86]
Statistical Analysis 2: Comparison: Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib vs Cohort 1 and 2: Capecitabine; This Statistical Analysis corresponds to Nausea and vomiting scale; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.45 to 0.76]
Statistical Analysis 3: Comparison: Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib vs Cohort 1 and 2: Capecitabine; This Statistical Analysis corresponds to Pain scale; Test type: Superiority; p = 0.042, Regression, Cox; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.62 to 0.99]
Statistical Analysis 4: Comparison: Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib vs Cohort 1 and 2: Capecitabine; This Statistical Analysis corresponds to Dyspnea scale; Test type: Superiority; p = 0.599, Regression, Cox; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.81 to 1.44]
Statistical Analysis 5: Comparison: Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib vs Cohort 1 and 2: Capecitabine; This Statistical Analysis corresponds to Insomnia scale; Test type: Superiority; p = 0.196, Regression, Cox; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.64 to 1.10]
Statistical Analysis 6: Comparison: Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib vs Cohort 1 and 2: Capecitabine; This Statistical Analysis corresponds to Appetite loss scale; Test type: Superiority; p = 0.011, Regression, Cox; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.54 to 0.92]
Statistical Analysis 7: Comparison: Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib vs Cohort 1 and 2: Capecitabine; This Statistical Analysis corresponds to Constipation scale; Test type: Superiority; p = 0.564, Regression, Cox; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.83 to 1.41]
Statistical Analysis 8: Comparison: Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib vs Cohort 1 and 2: Capecitabine; This Statistical Analysis corresponds to Diarrhea scale; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.32 to 0.55]
Statistical Analysis 9: Comparison: Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib vs Cohort 1 and 2: Capecitabine; This Statistical Analysis corresponds to Financial difficulties scale; Test type: Superiority; p = 0.118, Regression, Cox; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.56 to 1.07]

16. Secondary Outcome: Time to Deterioration (TTD) in EORTC QLQ-BR23 Functional Scale
Description: Time to deterioration is defined as the time from the date of randomization to the date of first detection of deterioration for QLQ-BR23 score [(date of first detection of deterioration - date of randomization + 1). Deterioration is defined as a change from baseline ≥ minimally important difference (MID) for QLQ-BR23 score. Patients without deterioration have been censored at their last quality of life assessment. For patients with no post-baseline assessment time to deterioration have been censored at Day 1.
  Sexual functioning and Sexual enjoyment could not be estimated due to lack of response.
  999 means value not estimated.
Time Frame: as for outcome 8
Population: QoL population: a subset of enrolled patients with available QoL questionnaires (the baseline and at least one more).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib | Cohort 1 and 2: Capecitabine
Number analyzed (Participants) | 268 | 269
months
  Body image | 8.1 [5.6 to 9.3] | 7 [4.7 to 11.8]
  Future perspective | 28.1 [14.3 to NA] — Insufficient number of participants with events | 47.8 [25.1 to 47.8]
Statistical Analysis 1: Comparison: Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib vs Cohort 1 and 2: Capecitabine; This Statistical Analysis corresponds to Body image scale; Test type: Superiority; p = 0.659, Regression, Cox; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.74 to 1.21]
Statistical Analysis 2: Comparison: Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib vs Cohort 1 and 2: Capecitabine; This Statistical Analysis corresponds to Future perspective scale; Test type: Superiority; p = 0.928, Regression, Cox; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.74 to 1.39]

17. Secondary Outcome: Time to Deterioration (TTD) in EORTC QLQ-BR23 Symptom Scale
Description: Time to deterioration is defined as the time from the date of randomization to the date of first detection of deterioration for QLQ-BR23 score [(date of first detection of deterioration - date of randomization + 1). Deterioration is defined as a change from baseline ≥ minimally important difference (MID) for QLQ-BR23 score. Patients without deterioration have been censored at their last quality of life assessment. For patients with no post-baseline assessment time to deterioration have been censored at Day 1.
  Upset by hair loss could not be estimated due to lack of response.
Time Frame: as for outcome 8
Population: QoL population: a subset of enrolled patients with available QoL questionnaires (the baseline and at least one more).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib | Cohort 1 and 2: Capecitabine
Number analyzed (Participants) | 268 | 269
months
  Systemic side-effects | 4 [3.7 to 5.6] | 3.3 [2.8 to 4.3]
  Breast symptoms | 11.1 [9.3 to 16.7] | 11.5 [8.6 to 17.7]
  Arm symptoms | 8.8 [5.9 to 15] | 8.3 [4.9 to 13.4]
Statistical Analysis 1: Comparison: Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib vs Cohort 1 and 2: Capecitabine; This Statistical Analysis corresponds to Systemic side-effects scale; Test type: Superiority; p = 0.029, Regression, Cox; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.64 to 0.98]
Statistical Analysis 2: Comparison: Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib vs Cohort 1 and 2: Capecitabine; This Statistical Analysis corresponds to Breast symptoms scale; Test type: Superiority; p = 0.571, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.71 to 1.21]
Statistical Analysis 3: Comparison: Cohort 1 and 2: (Exemestane or Fulvestrant) Plus Palbociclib vs Cohort 1 and 2: Capecitabine; This Statistical Analysis corresponds to Arm symptoms scale; Test type: Superiority; p = 0.187, Regression, Cox; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.66 to 1.09]

ADVERSE EVENTS:
Time Frame: Through study treatment, an average of 8 months. All-Cause Mortality, through study treatment and follow up to approximately 34 months.
Description: AE were reported after Informed Consent Document (ICD) and before study drugs until approximately 30 days following the discontinuation of study treatment.
  All-Cause Mortality were reported from randomization until death (up to approximately 34 months).
Groups:
- Cohort 1: Palbociclib Plus Exemestane: Cohort 1:Palbociclib 125 mg orally once daily on Day 1 to Day 21 followed by 7 days off treatment on every 28 days cycles in combination with Exemestane 25 mg orally once daily.
  Palbociclib
  Exemestane
Arm/Group | Cohort 1: Palbociclib Plus Exemestane | Cohort 2: Palbociclib Plus Fulvestrant | Cohort 1 and 2: Capecitabine
All-Cause Mortality (participants affected / at risk) | 85/150 | 43/149 | 116/289
Serious Adverse Events (participants affected / at risk) | 34/150 | 21/149 | 72/289
Other Adverse Events (participants affected / at risk) | 147/150 | 148/149 | 286/289
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Palbociclib Plus Exemestane (N=150) | Cohort 2: Palbociclib Plus Fulvestrant (N=149) | Cohort 1 and 2: Capecitabine (N=289)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 1
Bone fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Breast infection (Infections and infestations) | 0 | 1 | 0
Bronchial infection (Infections and infestations) | 0 | 1 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 16
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 3
Fever (General disorders) | 1 | 1 | 2
Gallbladder infection (Infections and infestations) | 0 | 1 | 0
Ileitis (Gastrointestinal disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Heart failure (Cardiac disorders) | 1 | 1 | 1
Hematoma (Vascular disorders) | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Bacteremia (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 4
Respiratory infection (Infections and infestations) | 3 | 4 | 3
Dislocation of hip (Injury, poisoning and procedural complications) | 0 | 1 | 0
Drug overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ischemia cerebrovascular (Nervous system disorders) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1
Lymphedema (Vascular disorders) | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1
Mucositis (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 1
Chronic myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Urinary bladder carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 2
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2
Platelet count decreased (Blood and lymphatic system disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 2 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Stroke (Nervous system disorders) | 1 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Hip replacement (Surgical and medical procedures) | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 7
Tooth infection (Infections and infestations) | 1 | 0 | 0
Typhlitis (Gastrointestinal disorders) | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 2 | 1
Uveitis (Eye disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Palbociclib Plus Exemestane (N=150) | Cohort 2: Palbociclib Plus Fulvestrant (N=149) | Cohort 1 and 2: Capecitabine (N=289)
Fatigue (General disorders) | 83 | 76 | 169
Neutrophil count decreased (Blood and lymphatic system disorders) | 94 | 94 | 41
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 | 2 | 210
Diarrhea (Gastrointestinal disorders) | 30 | 26 | 161
Hypertension (Vascular disorders) | 51 | 55 | 111
Nausea (Gastrointestinal disorders) | 36 | 37 | 109
Mucositis (Skin and subcutaneous tissue disorders) | 40 | 25 | 87
Weight loss (Investigations) | 29 | 34 | 76
Vomiting (Gastrointestinal disorders) | 27 | 23 | 84
Weight gain (Investigations) | 33 | 24 | 74
Anorexia (Metabolism and nutrition disorders) | 23 | 18 | 68
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 28 | 49
Hypothermia (General disorders) | 28 | 20 | 45
Headache (Nervous system disorders) | 25 | 26 | 38
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 29 | 17 | 39
Constipation (Gastrointestinal disorders) | 23 | 14 | 42
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 19 | 26
Nail disorder (Skin and subcutaneous tissue disorders) | 7 | 4 | 58
Abdominal pain (Gastrointestinal disorders) | 17 | 4 | 43
Dizziness (Nervous system disorders) | 12 | 11 | 39
Dyspepsia (Gastrointestinal disorders) | 18 | 10 | 32
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 16 | 22
Fever (General disorders) | 16 | 12 | 29
Pruritus (Skin and subcutaneous tissue disorders) | 23 | 11 | 23
Obesity (Metabolism and nutrition disorders) | 12 | 15 | 28
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 14 | 29
Bone pain (Musculoskeletal and connective tissue disorders) | 18 | 11 | 25
Anemia (Blood and lymphatic system disorders) | 9 | 17 | 26
Flu like symptoms (General disorders) | 15 | 15 | 20
Dysgeusia (Nervous system disorders) | 9 | 7 | 29
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 18 | 11
Pain (General disorders) | 15 | 8 | 18
Hot flashes (Vascular disorders) | 15 | 10 | 2

LIMITATIONS AND CAVEATS:
Potential limitations of the study are:

* capecitabine outcome was better than that initially anticipated (9 months compared with 6 months in the protocol assumptions)
* open-label study design may lead to biased interpretations
* the subtype classification for the exploratory objective was carried out in 70% of patients in the primary tumour, which might have changed in the metastatic disease in a proportion of patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 30 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor can require changes to the communication.

DOCUMENTS (2):
  • Study Protocol (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT02028507/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/07/NCT02028507/SAP_001.pdf